CLINICAL TRIAL: NCT06933511
Title: The Impact of Diabetic Polyneuropathy on Shear Wave Elastography, Ultrasonographic Findings, and Hand Function in Carpal Tunnel Syndrome
Brief Title: Impact of Diabetic Polyneuropathy on Carpal Tunnel Syndrome: Shear Wave Elastography, Ultrasound, and Hand Function
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Burcu Sevingül, Medical Doctor (Physical Medicine and Rehabilitation Resident Doctor), Ankara Etlik City Hospital
Other Study IDs: AESH-BSevingul-02-003
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Carpal Tunnel Syndrome (CTS); Diabetic Polyneuropathy; Shear Wave Elastography; Median Nerve; Ultrasound; Hand Function
Keywords: Carpal Tunnel Syndrome; Diabetic Polyneuropathy; Shear wave elastography; Ultrasound; Median nerve; hand function
MeSH Terms: conditions — Carpal Tunnel Syndrome; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- (DM- / DPN- / CTS-): This group will serve as the control for the non-diabetic (DM-) patients with CTS and will be used to observe the effects of CTS alone. Additionally, it will serve as the control for the diabetic (DM+) patients without CTS and will be used to evaluate the effects of diabetes alone on the median nerve. In these patients, diagnoses of DPN and CTS will be excluded through electrodiagnostic testing.
- (DM- / DPN- / CTS+): The non-diabetic group with carpal tunnel syndrome (CTS) includes patients diagnosed with mild to moderate CTS through nerve conduction studies.
- (DM+ / DPN- / CTS-): The control group consists of diabetic (DM+) patients who have been excluded from diagnoses of diabetic polyneuropathy (DPN) and carpal tunnel syndrome (CTS) based on electrodiagnostic tests.
- (DM+ / DPN- / CTS+): The diabetic group with carpal tunnel syndrome (CTS) but without diabetic polyneuropathy (DPN) includes patients who were diagnosed with mild to moderate CTS and excluded from having DPN, both based on nerve conduction studies.
- (DM+ / DPN+ / CTS-): The diabetic group with diabetic polyneuropathy (DPN) but without carpal tunnel syndrome (CTS) includes patients who were diagnosed with DPN and excluded from having CTS, both based on nerve conduction studies.
- (DM+ / DPN+ / CTS+): The diabetic group with carpal tunnel syndrome (CTS) and diabetic polyneuropathy (DPN) includes patients diagnosed with mild to moderate CTS and DPN, both based on nerve conduction studies.

SUMMARY:
This observational study examines changes in the median nerve in patients diagnosed with diabetic polyneuropathy (DPN) and carpal tunnel syndrome (CTS) using shear wave elastography, microvascular imaging, and cross-sectional area measurements. It also compares the individual and combined effects of type 2 diabetes mellitus, DPN, and CTS on symptoms and hand function.

DETAILED DESCRIPTION:
After giving written consent, all participants will undergo a screening process to determine if they meet the eligibility criteria for the study. Those who qualify will proceed to the assessment phase.

In the physical examination, participants will undergo several tests on both hands, including Tinel's sign, Phalen's test, joint position sense, two-point discrimination (using a Baseline aesthesiometer), sensory assessment of light touch, hand grip strength (measured with a Baseline hand dynamometer), precision grips (tip-to-tip, lateral, and three-finger grip using a pinch meter), and fine manual dexterity (assessed using the Nine-Hole Peg Test). The distribution of symptoms will be evaluated using the Katz Hand Diagram. Symptom severity will be assessed with the Visual Analog Scale (VAS), the Boston Carpal Tunnel Questionnaire (BCTQ), and the Toronto Clinical Scoring System (TCSS). Disability in the upper extremity will be measured with the Quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH) questionnaire.

All participants will undergo ultrasound examination of the median nerve, including cross-sectional area (CSA) measurements and shear wave elastography (SWE) at the wrist (pisiform-scaphoid bone landmarks) and 12 cm proximal to the wrist. We will perform microvascular imaging (MVI) grading at the wrist. We will use the General Electric (GE) LOGIQ Fortis ultrasound device to measure CSA, MVI, and SWE. We will use two different transducers based on the measurement type: the L6-24 'hockey stick' transducer (22 MHz) for CSA and MVI, and the L2-9 linear transducer (14-8 MHz) for SWE assessments.

Following the ultrasound, participants will undergo electrodiagnostic evaluations on all four limbs, which will include sensory and motor conduction studies. Sensory conduction studies will include median nerve stimulation at the wrist with recordings taken from the second digit, and ulnar nerve stimulation at the wrist with recordings from the fifth digit. Additionally, the sensory distal latency difference between the median and ulnar nerves will be assessed by recording from the fourth digit. Motor conduction studies will involve median nerve stimulation at the wrist and antecubital fossa, with recordings from the abductor pollicis brevis muscle. Ulnar nerve conduction will be assessed by stimulating at the wrist, above and below the elbow, with recordings from the abductor digiti minimi. For the lower extremities, the peroneal nerve will be stimulated at the anterior ankle, below the fibular neck, and at the lateral popliteal fossa, with recordings taken from the extensor digitorum brevis. The tibial nerve will be stimulated at the posterior medial malleolus and popliteal fossa, with recordings from the abductor hallucis. The sural sensory conduction study will be performed by stimulating between the heads of the gastrocnemius muscle and recording from the posterior lateral malleolus. In addition, F-wave latency and sympathetic skin response will be measured for the early detection of diabetic polyneuropathy (DPN). In our laboratory, electrodiagnostic evaluations are routinely performed in accordance with the polyneuropathy protocol defined by Shin J. Oh. This protocol includes motor and sensory nerve conduction studies of the median nerve (motor: wrist to elbow; sensory: finger to wrist) in one upper extremity, as well as bilateral motor conduction studies of the posterior tibial and peroneal nerves, and bilateral sensory conduction studies of the sural nerves in the lower extremities. Polyneuropathy is defined as the presence of conduction slowing, reduced amplitude of the action potential, or absence of an evoked response in at least two nerves. Patients who meet this definition and also fulfill the American Association of Neuromuscular and Electrodiagnostic Medicine (AANEM) simplified criteria will be included in the study. According to the AANEM simplified criteria, a diagnosis of distal symmetric polyneuropathy can be made when abnormalities are detected in at least two nerves-one of which must be the sural nerve-across motor and/or sensory nerve conduction studies performed on a minimum of three limbs, including at least one lower extremity. Based on the electrophysiological classification of carpal tunnel syndrome (CTS) by Padua et al., patients with mild or moderate CTS will be included in the study. Mild CTS is characterized by a slowing of sensory conduction velocity in the median nerve, while distal motor latency remains within normal limits. Moderate CTS is defined by a slowing of median sensory conduction in the second digit-wrist segment, accompanied by an abnormal distal motor latency.

Data will be analyzed on a hand-by-hand basis. Based on G*Power analysis, each group will include at least nine hands. Hands will be categorized into six groups according to electrodiagnostic findings as follows: 1) No diabetes, no DPN, no CTS (DM- / DPN- / CTS-); 2) No diabetes, no DPN, with CTS (DM- / DPN- / CTS+); 3) With diabetes, no DPN, no CTS (DM+ / DPN- / CTS-); 4) With diabetes, no DPN, with CTS (DM+ / DPN- / CTS+); 5) With diabetes, with DPN, no CTS (DM+ / DPN+ / CTS-); and 6) With diabetes, with DPN, with CTS (DM+ / DPN+ / CTS+). These six groups will be compared in terms of ultrasound findings, symptoms, and hand function. The hypothesis being tested is based on the "double crush theory," which suggests that DPN may increase the susceptibility of the median nerve to entrapment, potentially making CTS more likely, and CTS may present as an early sign of DPN. The study will assess the combined effects of DPN and CTS on symptoms and hand function. We will also investigate how the presence of DPN, in addition to CTS, affects symptoms and hand function.

Our secondary objective is to investigate the effects of CTS on the median nerve in the population with DPN, by assessing CSA, MVI, SWE, symptoms, and hand function.

ELIGIBILITY:
Inclusion Criteria:

Patient Group:

* Presence of carpal tunnel syndrome (CTS) symptoms, including pain, numbness, tingling, burning, and weakness, which worsen during sleep, prolonged hand positions, or repetitive wrist movements, and improve with hand shaking or changing position.
* Cognitively able to understand and participate in the study.
* Aged between 18 and 78 years.
* Has given written informed consent to participate.

Control Group:

* Asymptomatic individuals, with or without diabetes.
* Cognitively able to understand and participate in the study.
* Aged between 18 and 78 years.
* Has given written informed consent to participate.

Exclusion Criteria:

* History of previous carpal tunnel surgery or injection.
* History of previous upper extremity trauma.
* Presence of mass lesions or any condition that compresses the median nerve, observed during ultrasonographic examination.
* Presence of a persistent median artery.
* Presence of a bifid or trifid median nerve.
* Presence of anastomoses, such as Martin-Gruber.
* History of long-term excessive alcohol consumption.
* Chronic renal failure.
* Presence of neuropathy due to a neurological condition.
* Thyroid disorders.
* History of malignancy.
* History of neurotoxic drug use.
* Peripheral arterial occlusive disease.
* Severe diabetic polyneuropathy (DPN) diagnosis.
* Pregnancy.
* Cervical radiculopathy or brachial plexopathy.
* Osteoarthritis of the hand.
* Rheumatologic disease.
* Systemic autoimmune disease.
* History of cerebrovascular disease.
* Dupuytren's contracture.
* Sclerodactyly.
* Cognitive limitations that would prevent understanding the study protocol.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include non-diabetic individuals, diabetic individuals with diabetic polyneuropathy (DPN), and diabetic individuals without diabetic polyneuropathy. Participants will be selected based on clinical presentation of hand symptoms such as pain, numbness, tingling, burning, and weakness, and each participant will be assessed for the presence or absence of carpal tunnel syndrome (CTS). Participants from both the diabetic and non-diabetic populations will be included in the study, with both CTS and non-CTS subgroups in each population.
Sampling Method: Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2025-04-18 (Estimated); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Sonographic and symptomatic assessment of median nerve | baseline (single session)
  This study investigates how diabetic polyneuropathy (DPN) affects the development and clinical signs of carpal tunnel syndrome (CTS). We will assess the median nerve by measuring its cross-sectional area (CSA), stiffness using shear wave elastography (SWE), and symptom severity with the Boston Carpal Tunnel Questionnaire (BCTQ). The BCTQ is a self-reported questionnaire with 11 items for symptom severity and 8 for functional impairment, each scored from 1 to 5. Higher scores reflect worse symptoms or greater disability. CSA will be measured three times within the median nerve's epineurium-both at the carpal tunnel entrance and on the forearm. SWE will also be measured at these locations, using three circular regions of interest (2-4 mm) selected from the most reliable areas shown on the reliability index map.

SECONDARY OUTCOMES:
Microvascular Imaging (MVI) of the Median Nerve | baseline (single session)
  To detect vascular changes in the median nerve associated with CTS and DPN using Doppler ultrasonography. Microvascular Imaging (MVI) was used instead of power Doppler ultrasound due to its superior ability to visualize small-diameter vessels and low blood flow. Microvascularity was graded into four categories: Grade 0 indicates no detectable blood flow; Grade 1 indicates 1-2 isolated flow signals; Grade 2 represents more than two flow points or 1-2 flow strips longer than 1 mm; and Grade 3 denotes more than three continuous flow strips.
Polyneuropathy Symptom Severity Using the Toronto Clinical Scoring System (TCSS) | baseline (single session)
  The Toronto Clinical Scoring System (TCSS) is a comprehensive assessment tool divided into three sections. The first section evaluates the presence of symptoms in both the upper and lower extremities, including pain, numbness, tingling, burning, weakness, and instability. A score of 1 is given for each symptom present and 0 for those absent. The second section evaluates reflexes by assessing patellar and Achilles reflexes on both sides. Reflexes are scored as 0 for normal, 1 for reduced, and 2 for absent. The third section involves sensory testing of the great toe, including pinprick, light touch, vibration, thermal sensation, and joint position sense, scoring 0 for normal and 1 for abnormal sensation. The TCSS provides a way to assess the severity of diabetic polyneuropathy and is also useful for monitoring disease progression or response to treatment.
Hand Function Evaluation with Grip Strength, Nine-Hole Peg Tests and Q-DASH Questionnaire | baseline (single session)
  The Quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH) questionnaire is a self-reported tool that assesses the impact of upper extremity disorders on daily activities, including symptoms and physical limitations. It consists of 11 items, with higher scores indicating greater disability and impairment in hand function. We will measure hand grip strength and test three types of precise grip strength: lateral pinch (similar to holding a key), tip-to-tip pinch (similar to holding a needle), and three-finger pinch (similar to holding a pen). For each type of grip, the average score will be recorded after one-minute intervals. The Nine-Hole Peg Test (NHPT) assesses fine motor skills, manual dexterity, and hand function, providing objective data on the speed and accuracy of hand movements, including for conditions such as carpal tunnel syndrome (CTS).

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Sevingul, M.D., Principal Investigator — Ankara Etlik City Hospital; Burcu Sevingul, M.D., Study Director — Ankara Etlik City Hospital; Ebru Karaca Umay, M.D., Study Chair — Ankara Etlik City Hospital; Alper Dilli, M.D., Study Chair — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Kim J, Kim MW, Kim JM. Enhanced diagnosis and severity assessment of carpal tunnel syndrome using combined shear wave elastography and cross-sectional area analysis: A prospective case-control study. PLoS One. 2025 Mar 24;20(3):e0320011. doi: 10.1371/journal.pone.0320011. eCollection 2025. PMID 40127092
- [Result] Martikkala L, Pemmari A, Himanen SL, Makela K. Median Nerve Shear Wave Elastography Is Associated With the Neurophysiological Severity of Carpal Tunnel Syndrome. J Ultrasound Med. 2024 Jul;43(7):1253-1263. doi: 10.1002/jum.16450. Epub 2024 Mar 22. PMID 38516753
- [Result] Sung JH, Kwon YJ, Baek SH, Son MH, Lee JH, Kim BJ. Utility of shear wave elastography and high-definition color for diagnosing carpal tunnel syndrome. Clin Neurophysiol. 2022 Mar;135:179-187. doi: 10.1016/j.clinph.2021.10.020. Epub 2021 Dec 10. PMID 34963555
- [Result] Wee TC, Simon NG. Shearwave Elastography in the Differentiation of Carpal Tunnel Syndrome Severity. PM R. 2020 Nov;12(11):1134-1139. doi: 10.1002/pmrj.12334. Epub 2020 Feb 14. PMID 31994817
- [Result] Park D, Lee SE, Cho JM, Yang JW, Kim M, Kwon HD. Characteristics of diabetic and non-diabetic carpal tunnel syndrome in terms of clinical, electrophysiological, and Sonographic features: a cross-sectional study. BMC Musculoskelet Disord. 2023 Sep 16;24(1):739. doi: 10.1186/s12891-023-06881-1. PMID 37716949